CLINICAL TRIAL: NCT06973941
Title: Effectiveness and Feasibility of Virtual Reality Relaxation Compared to Guided Imagery Relaxation in Older Adults With Mental Illness: A Randomized Controlled Study
Brief Title: VR Relaxation in Older Adults With Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Sandra Anna, Associate Professor, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 410522
Record Dates: First submitted 2025-05-06; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Mental Disorder
Keywords: relaxation; aging; virtual reality; mental health
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Prior to the relaxation exercise, the patients receive a short training session on how to wear the VR headset, for which Oculus Meta Quest 2 (Reality Labs, Meta Platforms Inc) is used, and on how to navigate in the virtual world. Patients are informed that the investigator would stay in the room during the relaxation exercise but would not actively interact with them until the 10-minute intervention was over (except if they needed assistance or wished to stop). After the investigator starts the VR relaxation application, which is part of the app "Nature Treks VR" by Greenergames (released on May 21, 2019), the patients put on the headset and proceed with the relaxation exercise. The virtual world is a natural environment providing a view of a forest with a nearby river, mountains in the distance, flowers and animals, accompanied by relaxing music and the sound of birds chirping. All patients experience the same relaxing environment.
  Interventions: Other: Virtual reality relaxation
- Guided Imagery (Active Comparator): Patients receive an audio guided dream journey, conducted by one of the investigators. The dream journey is exclusively developed for the purpose of this study by an experienced psychiatrist to ensure comparability and to control for familiarity, since this type of relaxation exercise is implemented in regular geriatric psychiatric care. Duration (10 minutes in total) and content (forest, natural environment) of the GI-based dream journey are tailored as precisely as possible to the relaxing VR application. Thus, the dream journey describes a similar natural scene taking place in a forest with a river, flowers and animals in the surrounding area and mountains in the distance, accompanied by relaxing music and nature sounds. We ensure to only include specific elements, e.g. deers and rabbits, that are also visible in the VR environment and avoid any additional instructions not provided in the VR application.
  Interventions: Other: Guided imagery relaxation

INTERVENTIONS:
Other: Virtual reality relaxation — 10-minute VR relaxation application, part of the app "Nature Treks VR" by Greenergames (released on May 21, 2019), used with a Metaquest head-mounted display
  Arms: Virtual Reality
Other: Guided imagery relaxation — 10-minute guided imagery relaxation where an investigator reads a dream journey
  Arms: Guided Imagery

SUMMARY:
This clinical trial is exploring whether virtual reality (VR) can be a helpful and practical tool for reducing stress and anxiety in older adults receiving mental health care. The study compares two common relaxation methods: one using traditional guided imagery (a technique that uses calming mental pictures) and one using immersive VR technology.

Participants are older adults with mental health conditions who take part in a single relaxation session using either VR or guided imagery. Before and after the session, researchers measure how relaxed, calm, and emotionally well the participants feel.

The study aims to answer several questions:

Do both methods reduce anxiety and negative emotions right after the session?

Do they increase relaxation, well-being, and positive feelings?

Is VR more effective than guided imagery for this group?

Does feeling more immersed in the VR environment lead to lower anxiety?

Researchers are also evaluating whether these techniques are comfortable and practical for older adults by looking at factors like satisfaction, drop-out rates, and ease of use.

Because relaxation exercises are already used in older adult mental health care, this research could help improve how such techniques are delivered - especially if VR turns out to be a powerful, accessible option for this population.

DETAILED DESCRIPTION:
This single-blinded pilot randomized controlled trial investigates the effectiveness and feasibility of virtual reality (VR)-based relaxation compared to guided imagery (GI)-based relaxation among older adults receiving inpatient psychiatric care. The study targets geriatric patients with various mental health diagnoses to evaluate whether immersive VR experiences offer comparable or superior benefits to a traditional guided imagery intervention.

The primary objectives are to determine whether:

Both interventions lead to an immediate reduction in state anxiety, negative affect, and perceived stress.

Both interventions result in an immediate increase in well-being, positive affect, and perceived relaxation.

Participants in the VR group show greater improvements in psychological outcomes than those in the GI group.

In the VR group, a higher sense of presence predicts lower post-intervention state anxiety (the primary outcome).

Feasibility is assessed based on participant retention, self-reported satisfaction, overall experience, and-specifically for the VR group-motion sickness and sense of presence. The study hypothesizes that both interventions are feasible for this patient population, with minimal side effects and no significant influence of medical or sociodemographic factors on feasibility outcomes.

Design and Randomization:

Participants are randomly assigned in a 1:1 ratio to either the VR or GI condition using block randomization with a block size of four. Randomization is conducted using R Studio (version 4.4.2), ensuring balanced group allocation throughout the study. This method helps mitigate the impact of clinical setting variables, such as unplanned discharges, on group sizes.

Participant Procedures:

Following informed consent, each participant receives detailed information about the study, including its purpose, duration, and the voluntary nature of participation. Baseline data (T0) are collected via structured interviews and digital self-report questionnaires administered through REDCap on a tablet. If necessary, the investigator reads the questions aloud and records responses.

VR Group:

Participants allocated to the VR group complete a brief training on using the Oculus Meta Quest 2 headset. The intervention consists of a 10-minute immersive experience using the "Nature Treks VR" application, which features a calming natural environment with a forest, river, distant mountains, flowers, animals, and ambient nature sounds. All participants in this group view the same virtual environment to maintain standardization. The investigator remains in the room to offer assistance if needed but does not interact during the session unless requested.

GI Group:

Participants in the GI group listen to a 10-minute guided dream journey, designed specifically for this study by a psychiatrist. The audio script mirrors the VR environment, describing a peaceful forest scene with similar natural elements (e.g., deer, rabbits, river, mountains), accompanied by matching music and sounds. The script avoids additional guidance such as breathing cues to ensure comparability with the VR experience.

Post-Intervention Procedures:

Immediately after the session, participants in the VR group rate their experience of motion sickness. All participants then complete the post-intervention questionnaires (T1), consistent with their assigned condition. The full procedure lasts approximately 45 minutes for the VR group and 35 minutes for the GI group.

Outcomes:

Effectiveness is assessed at T0 and T1 using the State-Trait Anxiety Inventory, the Positive and Negative Affect Schedule, and Visual Analog Scales. Dropout rates, satisfaction and experience are compared. Motion sickness and sense of presence are measured with the Fast Motion Sickness Scale and the Igroup Presence Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* in psychiatric treatment at the St. Hedwig Hospital Berlin, Germany
* a psychiatric diagnosis (according to ICD-10)
* aged 55 years and older
* ability to understand the content of the study and provide written informed consent

Exclusion Criteria:

* insufficient proficiency in German language
* acute aggression
* acute suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
State anxiety | One pre- and post-intervention-measurement during a single session that takes 35-45 minutes.
  Assessed using the German version of the state subscale of the State-Trait Anxiety Inventory (STAI-X1; Laux et al., 1981; Spielberger et al., 1970), which has good psychometric properties, such as a high internal consistency (α = .90) (Laux et al., 1981). The STAI-X1 is a self-report questionnaire comprising 20 items in total, some of which need to be reversed. Short statements, such as 'I am nervous.' (indicating presence of anxiety) or 'I feel calm' (indicating absence of anxiety), had to be evaluated on a 4-point scale ranging from 1 = 'not at all' to 4 = 'very much'. Patients are asked to indicate to what extent each statement applied to them at that moment. A sum score between 20 and 80 iscalculated, with higher values indicating a higher level of state anxiety.

SECONDARY OUTCOMES:
Positive and negative affect | One pre- and post-intervention-measurement during a single session that takes 35-45 minutes.
  Evaluated with the German Version of the Positive and Negative Affect Schedule (PANAS; Breyer & Bluemke, 2016; Krohne et al., 1996; Watson et al., 1988). The PANAS is a 20 item self-report questionnaire assessing two dimensions of affect, positive affect (PA) and negative affect (NA), with 10 items for each dimension. Since it is allowed to adapt PANAS instructions depending on the research purpose (Breyer & Bluemke, 2016), we ask patients to refer to the present moment when evaluating each adjective on a 5-point Likert scale (1 = 'not at all' to 5 = 'extremely'). In a representative sample from the GESIS Panel 2014, the German version of the PANAS had good psychometric properties, such as high internal consistency (α = 0.86) (Breyer & Bluemke, 2016).
Perceived stress | One pre- and post-intervention-measurement during a single session that takes 35-45 minutes.
  Measured with a single-item VAS, which we developed for our study based on the Numeric Stress Rating Scale (NSRS; Lee, 2010, as cited in Tan et al., 2021). In an RCT on VR stress management for inpatients with mental disorders, the NSRS was used to assess immediate changes in subjective stress pre- and post-sessions. Test-retest reliability was indicated by significant correlations between waitlist control group scores (Tan et al., 2021). The VAS item was translated to German and adapted for the purpose of our study. Patients rate their momentary perceived stress on a scale from 0 = 'no stress' to 10 = 'extreme stress' (Tan et al., 2021). It is presented as a horizontal line with no calibration marks apart from the two labeled endpoints. Numeric mean scores for T0 and T1 are obtained, with lower scores indicating lower stress levels.
Perceived relaxation | One pre- and post-intervention-measurement during a single session that takes 35-45 minutes.
  Measured using a single-item VAS, which we developed and translated for this study based on previous studies examining the effects of VR relaxation in individuals with mental illness (Riches, Nicholson, et al., 2023; Tan et al., 2021). The patients are asked to mark on a scale how relaxed they feel at that moment. The scale ranges from 0 = 'not relaxed at all' to 10 = 'very relaxed' and is presented as a horizontal line with no calibration marks apart from the two labeled endpoints. Numeric mean scores for T0 and T1 are calculated, with higher scores indicating a higher momentary relaxation.
Overall well-being | One pre- and post-intervention-measurement during a single session that takes 35-45 minutes.
  Assessed using a single-item VAS. Patients are asked to mark on the VAS how well they feel at that present moment. The scale is presented as a horizontal line with two endpoints (0 = 'not well at all'; 10 = 'very well') and no marks along the scale. Numeric mean scores are calculated for T0 and T1, with higher values indicating a higher overall well-being.
Drop out rates | One measurement during a single session that takes 35-45 minutes.
  Drop-out rates are recorded to compare the acceptance of both treatments. Participants are considered as a drop-out, if the VR-based relaxation exercise or the guided dream journey is terminated before the scheduled end after 10 minutes.
Patients' satisfaction | One post-intervention-measurement during a single session that takes 35-45 minutes.
  Measured with five items, based on the ZUF-8 (Schmidt et al., 1989), which is the German version of the Client Satisfaction Questionnaire (CSQ-8; Attkisson & Zwick, 1982). The ZUF-8 is commonly used to economically evaluate patient's general satisfaction with psychotherapeutic treatment in stationary settings (Schmidt et al., 1989), but has already been adapted to examine the feasibility of VR relaxation in psychiatric outpatients (Humbert et al., 2023). For our study, three items are excluded due to their lack of suitability for our specific intervention context, five items are retained and slightly rephrased to adapt them to each condition. The response option for each item was adopted from the ZUF-8 (Schmidt et al., 1989).
Patients' experience | One post-intervention-measurement during a single session that takes 35-45 minutes.
  Assessed with three single-item VAS, ranging from 0 = 'not at all' to 10 = 'very'. The scales were adopted, partly rephrased and translated into German from the study of Riches, Nicholson, et al. (2023) on VR relaxation within acute psychiatric services. Patients rate how helpful they found the (virtual) relaxation exercise (helpfulness), how connected they felt to nature (connectedness to nature) and to what extent they felt that they were actually in the relaxing environment (immersion).
Motion Sickness | One post-intervention-measurement during a single VR session that takes 35-45 minutes.
  Measured as an indicator for the tolerability of the VR relaxation exercise, measured with the Fast Motion Sickness Scale (FMS; Keshavarz and Hecht, 2011), a valid and brief self-report measure to determine motion sickness in VR (Keshavarz & Hecht, 2011), immediately after the VR application was terminated. The patients rate the severity of their current motion sickness on a scale from 0 (no motion sickness) to 20 (frank motion sickness).
Sense of presence | One post-intervention-measurement during a single VR session that takes 35-45 minutes.
  Measured with the German version of the iGroup Presence Questionnaire (IPQ; Himmels et al., 2023). The IPQ has good psychometric properties (Himmels et al., 2023), was previously used to assess presence in VR-based relaxation interventions (Liszio et al., 2018), and demonstrated its feasibility for measuring sense of presence in a geriatric psychiatric sample (Just & Lütt et al., 2024). In total, 14 items are rated on a scale from -3 to +3, with varying anchors for each item. The IPQ items are divided into the subscales 'spatial presence,' 'involvement,' and 'realness,' with one additional item measuring 'general presence' (Himmels et al., 2023).

CONTACTS AND LOCATIONS:
Locations (1):
- Charité University Medicine, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Due to privacy and ethical considerations, individual-level data from this study cannot be shared publicly; however, reasonable requests will be reviewed within one week. We plan to openly share aggregated data relevant to the findings.